CLINICAL TRIAL: NCT05550792
Title: Cardiac Contractility Modulation in Patients With Chronic Heart Failure and the Various Forms of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Collaborators: Ministry of Health, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Alfiya Achatovna Safiullina, sub-Investigator, National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: КА-027-2018
Record Dates: First submitted 2022-01-26; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure; Atrial Fibrillation; Left Ventricular Ejection Fraction
Keywords: Cardiac contractility modulation; Atrial Fibrillation; Heart Failure; Narrow QRS Complex; left ventricular ejection fraction
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimizer device (Active Comparator): 100 patients were enrolled sequentially, 100 patients were implanted with an optimizer smart against the background of optimal drug therapy for heart failure
  100 patients were implanted with a CCM Optimizer device without an atrial lead, per the protocol specifications recived optimal drug therapy CHF The following studies were performed in the 100 patients with CHF and AF before implantation of the MCC device and after 2 and 6 и 12 months of follow-up: 12-channel ECG with an estimate of the width of the QRS complex, transthoracic EchoCG,Speckle-tracking EchoCG,Myocardial work, 6-minute walk test, determination of the level of Pro-natriuretic N-terminal peptide (NT-proBNP), Holter ECG, and a questionnaire based on the Minnesota quality of life questionnaire for patients with CHF (MHFLQ).
  Interventions: Device: optimizer smart
- Without Optimizer device (No Intervention): 100 patients were enrolled sequentially,100 patients received only optimal drug therapy for chronic heart failure 100 patients ( Without Optimizer device ) with CHF and AF before study and after 2 and 6 и 12 months of follow-up: 12-channel ECG with an estimate of the width of the QRS complex, transthoracic EchoCG,Speckle-tracking EchoCG,Myocardial work, 6-minute walk test, determination of the level of Pro-natriuretic N-terminal peptide (NT-proBNP), Holter ECG, and a questionnaire based on the Minnesota quality of life questionnaire for patients with CHF (MHFLQ).

INTERVENTIONS:
Device: optimizer smart — The CCM implantation procedure was performed in the right precordial region of the chest (the right subclavian area). Two active fixation Ingevity leads (Boston Scientific) were advanced via the right subclavian vein into the right ventricle (RV) and actively fixed to the right ventricular septum for ventricular sensing and delivery of CCM signals.
  Arms: Optimizer device

SUMMARY:
Chronic heart failure (CHF) is a global pandemic which affects around 26 million people worldwide and develops in 10% of people over 70 years . According to the results of the EPOCHA-CHF study, CHF is detected in 7-10% of cases in the Russian Federation . Atrial fibrillation (AF) is the most common arrhythmia in patients with both preserved (HFpEF) and reduced ejection fraction (HFrEF) heart failure. The prognostic impact of AF on CHF is negative, including the significant increase in mortality and hospitalization.

One of the common causes of decompensation of CHF is AF. The debut of AF in CHF is one of the markers of disease progression.

Rapid development in interventional cardiology due to the invention of cardiac catheter technologies during the last decades provided a new option for non-pharmacological treatment of CHF. Nowadays the use of electrophysiological methods of treatment can significantly improve the prognosis of CHF. Pacemakers, cardiac resynchronization devices, and cardioverter defibrillators are the most commonly implanted devices in patients with CHF.

In 2014, the European Society of Cardiology presented a report of the European Heart Rhythm Association on the use of new devices for CHF, including the Optimizer device for delivery of cardiac contractility modulation therapy (CCM) .

It is worth noting that CCM is a new step in the CHF treatment. This device is of proven benefit to patients with symptomatic heart failure on optimal medical therapy who do not qualify for cardiac resynchronization therapy.

Multiple studies of CCM show clinical improvement with this therapy, including metrics such as peak VO2, 6MW, and NYHA functional class. However, the vast majority of patients enrolled in these studies were patients in sinus rhythm.

As the technology progressed and the need for the trial sensing led wanted, further experiences incorporated patients with AF. A new generation of devices (Optimizer Smart®), which does not require the implantation of an atrial electrode made it possible to implant CCM in patients with AF.

The present trial demonstrates the results of a pilot study conducted in National Medical Research Center of Cardiology Ministry of Health of the Russian Federation which compares the efficacy of CCM in patients with AF and ischemic and non-ischemic CHF compared to patients who received only optimal drug therapy CHF

DETAILED DESCRIPTION:
Background: Chronic heart failure (CHF) and atrial fibrillation (AF) often coexist and lead to severe decompensation of patients' lifestyle. Nowadays device therapy such as cardiac contractility modulation (CCM), which is used in addition to medical treatment, can significantly impact further prognosis and outcomes of patients with such comorbidities.

Methods: In the National Medical Research Center of Cardiology we conducted a study dedicated to investigating the efficacy of CCM in patients with CHF and AF. 200 patients with Hf and AF were included in the study and were divided into two groups according to implantation of a heart contractility modulation device and optimal drug therapy. 100 patients were implanted with a CCM Optimizer device without an atrial lead, per the protocol specifications ( 1 group) and 100 patients ( 2 group) received only optimal drug therapy CHF The following studies were performed in the 200 patients with CHF and AF before implantation of the MCC device and after 2 and 6 и 12 months of follow-up: 12-channel ECG with an estimate of the width of the QRS complex, transthoracic EchoCG, Speckle-tracking EchoCG, Myocardial work, 6-minute walk test, determination of the level of Pro-natriuretic N-terminal peptide (NT-proBNP), Holter ECG, and a questionnaire based on the Minnesota quality of life questionnaire for patients with CHF (MHFLQ),Perfusion Single-Photon Emission Computed Tomography All patients received long-term optimal drug therapy for CHF before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Documented HFrEF (20-40%)
* NYHA FC II-III for at least 3 months before screening
* AF
* Optimal CHF therapy and the absence of decompensations in ≥ 1 month.

Exclusion Criteria:

* Refusal to participate in the study
* Placement on the heart transplant waiting list, or post heart transplantation
* Terminal CHF
* Co-morbid diseases that may adversely affect the safety and / or efficacy of treatment
* Recent surgical intervention or trauma
* Medical conditions that limit life expectancy to 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
cardiovascular death + hospitalization due to decompensation of HF | 12 month
  Number of Participants with cardiovascular death + hospitalization due to decompensation of HF

SECONDARY OUTCOMES:
death from all causes | 12 month
  Number of Participants with death from all causes
hospitalization for any reason | 12 month
  Number of Participants with hospitalization for any reason
development of AF paroxysm in patients with paroxysmal AF | 12 month
  Number of Participants with development of AF paroxysm in patients with paroxysmal AF
worsening of the course of CHF, which required an outpatient visit and increased doses of diuretics | 12 month
  Number of Participants with worsening of the course of CHF, which required an outpatient visit and increased doses of diuretics
complications that required removal of the MCC | 12 month
  Number of Participants with complications that required removal of the MCC

CONTACTS AND LOCATIONS:
Overall Officials: Alfiya Safiullina, phd, Principal Investigator — National Medical Research Center for Cardiology, Ministry of Health of Russian Federation
Locations (1):
- Alfiya Safiullina, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uskach TM, Safiullina AA, Sapel'nikov OV, Amanatova VA, Nikolaeva OA, Grishin IR, Nazarov BM, Tereshchenko SN. [Modulation of cardiac contractility in patients with chronic heart failure and atrial fibrillation]. Ter Arkh. 2020 Oct 14;92(9):8-14. doi: 10.26442/00403660.2020.09.000598. Russian. PMID 33346425
- [Result] Dobrovolskaya SV, Saidova MA, Safiullina AA, Uskach TM, Tereshchenko SN. [Evaluation of the effectiveness of the chronic heart failure therapy using the device cardiac contractility modulation according to the new non-invasive method of the myocardium work analysis]. Kardiologiia. 2021 Dec 31;61(12):31-40. doi: 10.18087/cardio.2021.12.n1849. Russian. PMID 35057719
- See also: Dynamics of Holter electrocardiogram monitoring in patients with chronic heart failure and atrial fibrillation on the background of cardiac contractility modulation — http://www.researchgate.net/publication/355310222_Dynamics_of_Holter_electrocardiogram_monitoring_in_patients_with_chronic_heart_failure_and_atrial_fibrillation_on_the_background_of_cardiac_contractility_modulation
- See also: The assessment of left ventricular myocardial work in patients with chronic heart failure receiving cardiac contractility modulation therapy — https://www.researchgate.net/publication/355371644_The_assessment_of_left_ventricular_myocardial_work_in_patients_with_chronic_heart_failure_receiving_cardiac_contractility_modulation_therapy
- See also: A comprehensive approach to the treatment of a patient with chronic heart failure with a reduced left ventricular ejection fraction — https://www.researchgate.net/publication/354401498_Kompleksnyj_podhod_k_leceniu_pacientki_s_hroniceskoj_serdecnoj_nedostatocnostu_so_snizennoj_frakciej_vybrosa_levogo_zeludocka
- See also: Implantation of a cardiac contractility modulator in chronic heart failure and atrial fibrillation: results of a 6-month follow-up of one hundred patients — https://www.researchgate.net/publication/350802972_Implantation_of_a_cardiac_contractility_modulator_in_chronic_heart_failure_and_atrial_fibrillation_results_of_a_6-month_follow-up_of_one_hundred_patients
- See also: Hibernating myocardium volume in patients with chronic ischemic heart failure under modulation of myocardial contractility — https://www.researchgate.net/publication/356395673_Hibernating_myocardium_volume_in_patients_with_chronic_ischemic_heart_failure_under_modulation_of_myocardial_contractility
- See also: Modulation of cardiac contractility in patients with chronic heart failure and atrial fibrillation — https://www.researchgate.net/publication/346215887_Modulation_of_cardiac_contractility_in_patients_with_chronic_heart_failure_and_atrial_fibrillation
- See also: P1491Cardiac contractility modulation in patients with chronic heart failure and atrial fibrillation: 6 months of follow-up — https://www.researchgate.net/publication/342268435_P1491Cardiac_contractility_modulation_in_patients_with_chronic_heart_failure_and_atrial_fibrillation_6_months_of_follow-up